CLINICAL TRIAL: NCT06313892
Title: The Effect of Synchronous Home Based Tele Exercise on Physical Function, Daily Physical Activity and Frailty in Dialysis Patients: A Randomized Pilot Trial
Brief Title: The Effect of Home Based Tel-Exercise on Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA24HD-2-05
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: End Stage Renal Disease; Hemodialysis Complication
Keywords: Inactivity; Tele exercise; Home based exercise; Hemodialysis; Frailty; Physical function
MeSH Terms: conditions — Kidney Failure, Chronic; Sedentary Behavior; Frailty

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Who Masked: Outcomes Assessor
Masking Description: A research project collaborator who is not informed about grouping of participants will obtain outcome measurements of the functional test. Outcome adjudicators, and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The participants in the study group will be given an online personalized exercise program at home in non dialysis days. Each session will be 40 to 45 min in duration for 3 days per week over 12 weeks, 36 sessions in total.
  Interventions: Behavioral: Home based Exercise
- Control group (No Intervention): Patients allocated to the control group will receive their standard nephrological care. Through the 12-week period, all control participants will be instructed to maintain the standard treatment regimen and to maintain their customary dietary and physical activity patterns.

INTERVENTIONS:
Behavioral: Home based Exercise — The participants in the study group will be given an online personalized exercise program at home in non dialysis days. Synchronous tele-exercise will be delivered using the free teleconference application (app) (Google Meets software). The groups of tele-exercises will be private and the professional will send the link for each training session and will control the access of the participants. Each session will be 40 to 45 min in duration for 3 days per week over 12 weeks, 36 sessions in total.
  Arms: Exercise group

SUMMARY:
The objective of the trial is to assess key areas of uncertainty regarding the use of synchronous home-based tele exercise in future practice and research, including issues relating to feasibility, safety and potential for efficacy.

DETAILED DESCRIPTION:
Patients with renal failure undergoing maintenance dialysis (HD) therapy typically have very low levels of physical activity (PA), and this is associated with greatly increased morbidity and mortality.

According to studies, regular exercise is beneficial for patients at all stages, and the current recommendations for the prevention and management of side effects in HD patients, especially in the elderly, is regular exercise because it improves physical performance and PA . Currently, due to the unfamiliarity of dialysis center staff and nephrologists with the benefits of exercise, only 10% of the world's clinics have a plan to exercise during HD. Therefore, home-based exercise programs are a suitable option for patients to reduce their costs and make it easy to adhere to.

Home-based exercise has the potential to utilize higher volume and higher intensity training if activity is monitored. However, many of these programs are unsupervised and this is one of the major disadvantages of home-based exercise programs. Lack of prior knowledge about the safety and benefits of exercise programs, fear of injury, and lack of interest or motivation are barriers to exercise at home.

Tele-rehabilitation is rehabilitation services provided to patients from distant locations using information and communication technologies.Several studies have reported the use of e health-based self-management interventions in chronic kidney disease patients.

However, further research is needed to better understand the extent to which these techniques are acceptable, safe and potentially effective for supporting individuals undergoing HD treatment, given their unique needs and risk profile, is unknown. Our study seeks to address this gap by conducting a pilot evaluation of synchronous home-based tele exercise intervention designed for HD patient.

ELIGIBILITY:
Inclusion Criteria:

1. being Aged 18 years and over
2. Regular in-center HD 3 times a week
3. completed at least 1 year of stable HD history
4. Without myocardial infarction within past 3 months
5. permission from their doctors
6. have decision making capacity to enable them to give informed consent to take part in the study
7. have access to a smart device (e.g. smart phone, laptop or tablet), and have internet access

Exclusion Criteria:

1) Unstable cardiac status (angina, decompensated congestive heart failure, severe arteriovenous stenosis, uncontrolled arrhythmias, etc.) 2) Active infection or acute medical illness 3) Hemodynamic instability 4) Labile glycemic control 5) Unable to exercise (lower extremity amputation with no prosthesis) 6) having severe musculoskeletal pain at rest or with minimal activity 7) Unable to sit, stand or walk unassisted (walking device such as cane or walker allowed) 8) Having shortness of breath at rest or with activities of daily living (NYHAClass IV) 9) individuals with exercise participation ≥ 3 times per week that addressed ≥ 2 of the domains 10) Unstable HD treatment and changing (titrating) medication regime 11) Excess inter-dialytic weight gain (>4 kg since last HD or exercise session) 12) Myocardial infarction within past 3 months

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 Month
  Determining recruitment by eligible number/enrolled number
Retention rates | 3 Months
  Determining retention rate by patients who completed visit 2 / recruited patients
Adherence rate | 3 Months
  Determining the adherence by the number of participation in exercise sessions by a participant / the number of the exercise sessions planned in the program

SECONDARY OUTCOMES:
Rate of changes of daily physical activity level | Pre test and 3 months later ( post test)
  To examine the effect of home-based synchronous tele-exercise on daily activity level by using Low Physical activity questionnaire.
  The questionnaire consists of 11 items that assess various parameters of physical activity within the past 7 days. These parameters include the amount of time spent walking around the neighborhood, for fitness or pleasure, and for transportation purposes, as well as the average duration of sedentary and sitting activities. The questionnaire also calculates the kilocalories expended during light, moderate, vigorous, and total physical activities.
Rate of changes of Frailty level | Pre test and 3 months later ( post test)
  To examine the effect of home-based synchronous tele-exercise on daily activity level by using Fried Frailty Index.
  Patients will be considered frail if they met 3 or more of the following 5 criteria: unintentional weight loss of 10 pounds or more in the prior year by self-report; exhaustion based on responses to two questions about energy; low physical activity based on the Minnesota questionnaire (< 383 kcal/wk for men or < 270 kcal/wk for women); slow gait speed (based on gender- and height-stratified cutoffs); and weak grip strength (based on gender- and BMI-stratified cutoffs). Patients will be asked whether they are independent in the following activities of daily living (ADLs): bathing, dressing, getting in and out of a chair, and walking around their home or apartment. Those reporting dependency in one or more will be considered to have an ADL limitation.
Rate of changes of physical function level | Pre test and 3 months later ( post test)
  To examine the effect of home-based synchronous tele-exercise on physical function level by 6 minute walk test and short physical performance battery test

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Study Director — Pardis Specialized Wellness Institute; Bobby Cheema, Dr, Principal Investigator — School of Health Sciences, Western Sydney University, Campbelltow, NSW 2560, Australia; Tomas Wilkinson, Dr, Principal Investigator — Diabetes Research Centre, University of Leicester, Leicester, UK; Kenneth Wilund, Dr, Principal Investigator — School of Nutritional Sciences and Wellness, Arizona University; Fabio Manferedini, Dr, Principal Investigator — Dept of Neuroscience and Rehabilitation, University of Ferrara
Locations (2):
- Iran (2):
  - Khorshid Dialysis Center, Isfahan
  - Pardis specialized wellness institute, Isfahan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the published article, after deidentification are to be shared
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Not applicable. It will be accessible for public.

REFERENCES:
- [Background] Rosa CS, Bueno DR, Souza GD, Gobbo LA, Freitas IF Jr, Sakkas GK, Monteiro HL. Factors associated with leisure-time physical activity among patients undergoing hemodialysis. BMC Nephrol. 2015 Nov 27;16:192. doi: 10.1186/s12882-015-0183-5. PMID 26613791
- [Background] Ortega-Perez de Villar L, Martinez-Olmos FJ, Perez-Dominguez FB, Benavent-Caballer V, Montanez-Aguilera FJ, Mercer T, Segura-Orti E. Comparison of intradialytic versus home-based exercise programs on physical functioning, physical activity level, adherence, and health-related quality of life: pilot study. Sci Rep. 2020 May 19;10(1):8302. doi: 10.1038/s41598-020-64372-y. PMID 32427935
- [Background] Manfredini F, Mallamaci F, D'Arrigo G, Baggetta R, Bolignano D, Torino C, Lamberti N, Bertoli S, Ciurlino D, Rocca-Rey L, Barilla A, Battaglia Y, Rapana RM, Zuccala A, Bonanno G, Fatuzzo P, Rapisarda F, Rastelli S, Fabrizi F, Messa P, De Paola L, Lombardi L, Cupisti A, Fuiano G, Lucisano G, Summaria C, Felisatti M, Pozzato E, Malagoni AM, Castellino P, Aucella F, Abd ElHafeez S, Provenzano PF, Tripepi G, Catizone L, Zoccali C. Exercise in Patients on Dialysis: A Multicenter, Randomized Clinical Trial. J Am Soc Nephrol. 2017 Apr;28(4):1259-1268. doi: 10.1681/ASN.2016030378. Epub 2016 Dec 1. PMID 27909047
- [Background] Knott S, Hollis A, Jimenez D, Dawson N, Mabbagu E, Beato M. Efficacy of Traditional Physical Therapy Versus Otago-Based Exercise in Fall Prevention for ALF-Residing Older Adults. J Geriatr Phys Ther. 2021 Oct-Dec 01;44(4):210-218. doi: 10.1519/JPT.0000000000000285. PMID 33534336
- [Result] Painter PL, Nelson-Worel JN, Hill MM, Thornbery DR, Shelp WR, Harrington AR, Weinstein AB. Effects of exercise training during hemodialysis. Nephron. 1986;43(2):87-92. doi: 10.1159/000183805. PMID 3713951
- [Result] Baggetta R, D'Arrigo G, Torino C, ElHafeez SA, Manfredini F, Mallamaci F, Zoccali C, Tripepi G; EXCITE Working group. Effect of a home based, low intensity, physical exercise program in older adults dialysis patients: a secondary analysis of the EXCITE trial. BMC Geriatr. 2018 Oct 20;18(1):248. doi: 10.1186/s12877-018-0938-5. PMID 30342464
- [Result] Hiraki K, Shibagaki Y, Izawa KP, Hotta C, Wakamiya A, Sakurada T, Yasuda T, Kimura K. Effects of home-based exercise on pre-dialysis chronic kidney disease patients: a randomized pilot and feasibility trial. BMC Nephrol. 2017 Jun 17;18(1):198. doi: 10.1186/s12882-017-0613-7. PMID 28623895
- [Result] Darawad MW, Khalil AA. Jordanian dialysis patients' perceived exercise benefits and barriers: a correlation study. Rehabil Nurs. 2013 Nov-Dec;38(6):315-22. doi: 10.1002/rnj.98. Epub 2013 May 23. PMID 23703743